CLINICAL TRIAL: NCT06652048
Title: High-dose Furmonertinib or Combined With Pemetrexed and Carboplatin/Cisplatin in EGFR-sensitive Mutation Advanced NSCLC After Disease Progression on First-line Treatment of Third-generation EGFR-TKI:a Multicencer,Open-label,Randomized Phase II Study
Brief Title: High-dose Furmonertinib or Combined With Chemotherapy in EGFR-mutant Advanced NSCLC After Disease Progression on Third-generation EGFR-TKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jialei Wang (Other)
Responsible Party: Sponsor-Investigator, Jialei Wang, Chief physician, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLAME-003-AST2818
Record Dates: First submitted 2024-10-10; First posted 2024-10-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Furmonertinib 160mg QD (Experimental): All patients enrolled into this group will receive furmonertinib 160mg p.o qd.
  Interventions: Drug: Furmonertinib 160mg QD
- Furmonertinib 240mg QD (Experimental): All patients enrolled into this group will receive furmonertinib 240mg p.o qd.
  Interventions: Drug: Furmonertinib 240mg QD
- Furmonertinib 160mg QD plus Chemotherapy (Experimental): All patients enrolled into this group will receive furmonertinib 160mg furmonertinib p.o qd plus chemotherapy[(carboplatin AUC 5 / cisplatin 75mg/m2+ pemetrexed 500mg/m2) every 21 days ×4 cycles + pemetrexed 500mg/m2 every 21 days maintenance]
  Interventions: Drug: Furmonertinib 160mg QD plus Chemotherapy

INTERVENTIONS:
Drug: Furmonertinib 160mg QD — All patients enrolled into this group will receive furmonertinib 160mg p.o qd.
  Arms: Furmonertinib 160mg QD
Drug: Furmonertinib 240mg QD — All patients enrolled into this group will receive furmonertinib 240mg p.o qd.
  Arms: Furmonertinib 240mg QD
Drug: Furmonertinib 160mg QD plus Chemotherapy — All patients enrolled into this group will receive furmonertinib 160mg furmonertinib p.o qd plus chemotherapy[(carboplatin AUC 5 / cisplatin 75mg/m2+ pemetrexed 500mg/m2) every 21 days ×4 cycles + pemetrexed 500mg/m2 every 21 days maintenance]
  Arms: Furmonertinib 160mg QD plus Chemotherapy

SUMMARY:
This is a multicenter, open-label,randomised phase II study planned to include 60 subjects with EGFR-sensitive mutation advanced NSCLC after disease progression on first-line treatment with third-generation EGFR-TKI.Eligible patients will randomly be assigned in a 1:1:1 ratio to receive 160mg/240mg furmonertinib p.o qd or 160mg furmonertinib p.o qd plus chemotherapy[(carboplatin AUC 5 / cisplatin 75mg/m2+ pemetrexed 500mg/m2) every 21 days ×4 cycles + pemetrexed 500mg/m2 every 21 days maintenance].Patients will be followed up every 2 cycles during the first half year , and every 3 cycles after the first half year.Treatment was continued until disease progression,intolerable toxic effects, investigator decision, patient withdrawal of consent, or death, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic non-small cell lung cancer ;
* Histologically or haematologically confirmed EGFR-sensitive mutations;
* Developed radiological progression after first-line third-generation EGFR-TKI monotherapy without any other subsequent systemic therapy. Patients received Osimertinib or Almonertinib for at least 3 months prior to progression and were discontinued 8 days prior to randomization, patients received Furmonertinib prior to progression achieved remission or sustained clinical benefit for at least 6 months (progression occurred during or <6 months after the last dose when the third-generation EGFR-TKI as a neoadjuvant/adjuvant , EGFR-TKI is considered as first-line treatment); Patients who had previously received chemotherapy or immunotherapy as neoadjuvant or adjuvant therapy could be included if they had metastatic/recurrent disease diagnosed more than 6 months after the last treatment and had radiographic progression after third-generation EGFR-TKI therapy;
* Patient has at least one accurately measurable lesion that has not been previously irradiated or biopsied during the screening period, according to RECIST 1.1; If the patient has one and only one measurable lesion, tissue biopsy of the lesion is permitted if the investigator assesses has limited impact on lesion detection, but baseline imaging of the lesion should be performed after tissue biopsy;
* Age ≥18 years old;
* ECOG 0-1 and had not worsened 2 weeks prior to enrollment;
* Life expectancy ≥ 12 weeks;
* Female patients of reproductive age must have a blood pregnancy test within 7 days before the first medication and it is negative; Infertile women can avoid pregnancy tests and contraception.;
* Able to comply with study protocols;
* Patient himself voluntarily participated and signed the informed consent.

Exclusion Criteria:

1. The tumor is confirmed by histology or cytology to be complicated with small cell lung cancer, neuroendocrine carcinoma, carcinosarcoma component or squamous cell carcinoma component exceeding 10%;
2. There are other driver gene mutations with known drug therapy (such as MET amplification, RET fusion, BRAF V600E mutation, etc.);
3. Allergy to the study drug and/or its excipients is known or suspected;
4. Treatment with any of the following:

   * Received any systemic anti-tumor therapy other than third-generation EGFR-TKI (including anti-tumor drugs in clinical research) before the first dose, and received cytotoxic drugs with significant delayed toxicity, such as mitomycin C and nitrosoureas, within 6 weeks before the first dose;
   * Received non-specific immunomodulators (including but not limited to interferon, IL-2), Chinese medicine or Chinese medicine preparations approved for anti-tumor indications within 2 weeks prior to initial administration;
   * Received a potent inhibitor of cytochrome P450 3A4 enzyme (CYP3A4) or a potent inducer within 7 days prior to the initial study drug administration, or who require continued treatment with these drugs during the study period;
   * Chest radiation therapy > 30 Gy within 6 months prior to initial dosing; Non-thoracic (except central nervous system) radiation therapy of >30 Gy within 4 weeks prior to initial dosing; Receiving palliative radiotherapy ≤30Gy within 2 weeks before the first dose;
   * Received intrapleural perfusion were not admitted until 28 days or more after the pleural fluid had stabilized;
   * Major surgery within 28 days of the first dose of study drug;
   * Patients with any factors that increase the risk of QTc prolongation or risk of Torsade ventricular tachycardia event who continuously take these medications during investigating period;
5. The toxicity associated with previous antitumor therapy did not return to ≤CTCAE Class 1, except for hair loss or chemotherapy-induced ≤CTCAE class 2 peripheral neurotoxicity;
6. There is spinal cord compression or symptomatic central nervous system (CNS) metastasis; Patients who were asymptomatic, stable, and did not require steroid treatment for 14 days or more before the first study drug administration were excluded. Patients who had received local CNS metastasis radiotherapy could only be enrolled after the end of radiotherapy and CNS metastasis symptoms were stable for 14 days or more;
7. Have other malignant tumors within the last 5 years or have a history of other malignant tumors, except skin basal cell carcinoma, cervical carcinoma in situ and breast ductal carcinoma in situ, which have been effectively controlled for more than 3 years;
8. Recent active peptic diseases, such as duodenal ulcer, ulcerative colitis, ileitis, etc., intestinal perforation, intestinal fistula, or other conditions that may lead to gastrointestinal bleeding or perforation as prescribed by the investigator; Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow study drugs, or prior major intestinal resection, which as determined by the investigator;
9. Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension, diabetes, and active bleeding, hepatitis B (Hepatitis B surface antigen (HBsAg) positive and HBV-DNA≥500 Active infections including IU/mL or higher than the lower limit of detection）, hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of detection), and human immunodeficiency virus (HIV) (including any patient receiving intravenous treatment for infection);
10. Past or current interstitial lung disease (ILD) or suspected ILD that could not be ruled out by imaging examination during screening;
11. Pulmonary complications resulting in clinically severe lung damage include, but are not limited to the following: Any serious underlying lung disease (e.g., pulmonary embolism diagnosed within 3 months prior to first dosing, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, etc.) b. Any autoimmune, connective tissue, or inflammatory diseases that may involve the lungs (such as rheumatoid arthritis, Sjogren's syndrome, and sarcoidosis), and other conditions that the investigator determines may increase the risk of developing interstitial pneumonia;
12. Any evidence of known corneal injury;
13. Examination within 28 days prior to administration of the first investigational drug revealed a lack of adequate bone marrow reserve or organ function；
14. Any condition meets the following cardiac standard:

    * Mean resting corrected QT interval (QTc)>470 msec, obtained from 3 ECG, using the screening clinic ECG machine-derived QTc value.
    * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block；
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
    * Echocardiographic examination: LVEF<50%，history of myocardial infarction, severe or unstable angina pectoris, coronary artery bypass surgery, or cardiac insufficiency ≥ NYHA Level 2 within the last 6 months；
15. Patients determined by the investigator to be unable to participate in the study, such as patients with a high probability of failing to comply with the study regulations, constraints, and requirements; Or other circumstances at the discretion of the investigator;
16. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival (PFS) assessed by INV per RECIST v1.1 in the FAS population.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Analysis will occur when PFS maturity is observed at approximately 12 months from the first patient begin study treatment
Objective Response Rate(ORR) | Up to 2 years
  Efficacy measures such as overall response rate (ORR), which is the proportion of subjects with CR or PR by INV based on RECIST v1.1
Duration of Response (DoR) | Up to 2 years
  Duration of response (DoR), which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival（OS） | Up to 2 years
  Overall Survival (OS) in the FAS population
Time to Subsequent Therapy (TTST) | Up to 2 years
  TTST is defined as the time from the date of randomization to the start date of the subsequent anti-cancer therapy following study treatment discontinuation, or death whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university shanghai cancer center, Shanghai, Shanghai Municipality, China